CLINICAL TRIAL: NCT05076903
Title: Effect of Opioid Free Anesthesia in Patients Undergoing Laparoscopic Gastrectomy: Subgroup Analysis Based on Psychological Trait
Brief Title: Effect of OFA in Laparoscopic Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Young Song, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3-2021-0295
Record Dates: First submitted 2021-09-05; First posted 2021-10-13 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients don't know which group they belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OFA group (Experimental): Dexmedetomidine and lidocaine are administered during anesthesia, and opioid is not used. For induction, 1 μg/kg of Dexmedetomidine is administered over 10 minutes and 1mg/kg of lidocaine is administered intavenously (bolus). This is followed by continuous intravenous infusion of dexmedetomidine at a rate of 0.2-0.7 μg/kg/h and infusion of lidocaine at the rate of 1 mg/kg/h.
  Interventions: Drug: OFA
- Control group (Active Comparator): Remifentanil is infused during anesthesia, and target-controlled infusion (TCI) is performed according to the Minto model. During indcution of anestheisa, target concentration of remifentanil is set within 3-5 ng/mL. After intubation, target concentration is adjusted within the range of 2-8 ng/mL.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: OFA — Dexmedetomidine and lidocaine are administered during anesthesia, and opioid is not used. For induction, 1 μg/kg of Dexmedetomidine is administered over 10 minutes and 1mg/kg of lidocaine is administered intavenously (bolus). This is followed by continuous intravenous infusion of dexmedetomidine at a rate of 0.2-0.7 μg/kg/h and infusion of lidocaine at the rate of 1 mg/kg/h.
  Arms: OFA group
Drug: Control — Remifentanil is infused during anesthesia, and target-controlled infusion (TCI) is performed according to the Minto model. During indcution of anestheisa, target concentration of remifentanil is set within 3-5 ng/mL. After intubation, target concentration is adjusted within the range of 2-8 ng/mL.
  Arms: Control group

SUMMARY:
The investigator will examine the effects of opioid free anesthesia in patients undergoing laparoscopic gastrectomy. The investigator expect that opioid free anesthesia will reduce postoperative pain and opioid consumption.

And investigator will analyze the association between postoperative pain and patient's underlying psychological characteristics and pain sensitivity. The investigator anticipate that psychological characteristics and pain sensitivity may be realted to postoperative pain and opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 19 years who underwent laparoscopic gastrectomy for gastric cancer

Exclusion Criteria:

* Patients with a history of allergic reactions to drugs
* Patients with a history of drug addiction
* Patients with chronic pain who require analgesics
* Patients with cancer other than the stomach
* History of hospitalization for psychiatric disorders
* Patients with sleep apnea
* Preoperative pulse oximetry (SpO2) < 95 %
* Moderate or severe hepatic impairment
* bradycardia (HR<50bpm), hypotension, atrioventricular block, intraventricular or sinus block
* Body mass index over 35 kg/m2
* Blood clotting disorders
* Pregnant/lactating women
* Cognitive impairment
* Unable to read consent form (eg illiterate, foreigner, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Opioid consumption in postoperative 24hrs | 24 hours after surgery
  Total opioid dose administered to the patient.

SECONDARY OUTCOMES:
Opioid consumption | postoperative 6hours, 12hours, 36hours, 48hours, 3days, 4days, 5days
  Total opioid dose administered to the patient.
Time to bowel function recovery (Gas passing time, Fluid intake start time, Soft diet start time) | up to 2weeks
  Time (hours) to first gas passing / starting oral fluid intake / starting soft diet
Pain score | postoperative 6hours, 12hours, 24hours, 36hours, 48hours, 3days, 4days, 5days, 2weeks
  verbal numerical rating scale 0-10
Nausea score | postoperative 6hours, 12hours, 24hours, 36hours, 48hours, 3days, 4days, 5days
  verbal numerical rating scale 0-10
Time to rescue analgesics after surgery | up to 2weeks
  Time (hours) to first rescue analgesics
Number of vomiting, antiemetic adeministration | up to 2weeks
  Number of vomiting, antiemetic adeministration
Hemodynamics during surgery | during surgery
  changes in hemodyanamics during surgery
QoR-15 | 1-5 days before surgery, postoperative 1day, postoperative 4day
  Score of QoR-15 questionnaire (Quality of Recovery-15)(Minimum value: 0, Maximum value: 150, higher scores means better.)
PCL-5 | postoperative 1week
  Score of PCL-5 (Posttraumatic stress disorder Checklist for DSM-5) (Minimum value: 0, Maximum value: 80, higher scores means worse.)

OTHER OUTCOMES:
Hospital Anxiety Depression Scale | 1-5 days before surgery
  Score of HADS questionnaire (Hospital Anxiety Depression Scale). It consists of 14 items and each item is scored on a scale of 0-3.
Euro Quality of Life - 5 Dimensions | 1-5 days before surgery
  Score of EQ-5D-5L questionnaire (Five-level version of Euro Quality of Life - 5 Dimensions). It consists of 5 items, and each item is scored on a scale of 1-5.
Patient Health Questionnaire | 1-5 days before surgery
  Score of PHQ-15 questionnaire (Patient Health Questionnaire-15). It consists of 15 items, and each item is scored on a scale of 0-2.
Pain Catastrophizing Scale | 1-5 days before surgery
  Score of PCS questionnaire (Pain Catastrophizing Scale). It consists of 13 items, and each item is scored on a scale of 0-4.
Big Five Inventory-10 | 1-5 days before surgery
  Score of BFI-10 questionnaire (Big Five Inventory-10). It consists of 10 items, and each item is scored on a scale of 1-5.
Hamilton Depression Rating Scale | 1-5 days before surgery
  Score of HAM-D (Hamilton Depression Rating Scale) examination. It consists of 17 items to evalulate depression, and higher scores indicate more severe depression.
Hamilton Anxiety Rating Scale | 1-5 days before surgery
  Score of HAM-A (Hamilton Anxiety Rating Scale) examination. It consists of 14 items to evalulate anxiety, and higher scores indicate more severe anxiety.
PainDETECT | 1-5 days before surgery
  Score of PainDETECT questionnaire. It consists of items such as the quality of pain, the pattern of pain, and higher scores indicate more severe neuropathic pain.
Temporal pain summation | 1-5 days before surgery
  Compare the pain after a single stimulation with the pain after 10 repeated stimulations.
Pressure pain threshold | 1-5 days before surgery
  The lowest pressure at which the participant perceives pain. It is measured by pressure algometry.
Pressure pain tolerance | 1-5 days before surgery
  The highest pressure when the participant perceived untolerable pain. It is measured by pressure algometry.
Frontal Electroencephalogram | perioperative period
  Band power and connectivity in electroencephalogram
Analgesia Nociception Index (ANI) | perioperative period
  Analgesia Nociception Index (ANI) from ANI monitoring

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Gangnam Severance Hospital, Seoul
  - Gangnam Severance Hsopital, Seoul

REFERENCES:
- [Derived] Bae MI, Oh J, Lee HS, Park S, Kwon IG, Song Y. Influence of psychological factors and pain sensitivity on the efficacy of opioid-free anesthesia: A randomized clinical trial. Gen Hosp Psychiatry. 2024 Jul-Aug;89:84-92. doi: 10.1016/j.genhosppsych.2024.04.001. Epub 2024 Apr 4. PMID 38838608